CLINICAL TRIAL: NCT03733717
Title: An Open-label, Multi-center Study to Evaluate the Pharmacokinetics, Safety, and Preliminary Efficacy of Isatuximab in Chinese Patients With Relapsed and/or Refractory Multiple Myeloma
Brief Title: Evaluation of Pharmacokinetics, Safety, and Preliminary Efficacy of Isatuximab in Chinese Patients With Relapsed and/or Refractory Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TED15085; U1111-1195-6028 (Other: UTN)
Record Dates: First submitted 2018-10-31; First posted 2018-11-07 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Multiple Myeloma
Keywords: Anti-CD38 monoclonal antibody
MeSH Terms: conditions — Multiple Myeloma | interventions — isatuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Isatuximab (Experimental): Administered intravenously every week in Cycle 1 (4 weeks) followed by every 2 weeks (Q2W) in subsequent cycles.
  Interventions: Drug: Isatuximab SAR650984

INTERVENTIONS:
Drug: Isatuximab SAR650984 — Pharmaceutical form: Concentrate for solution
  Route of administration: Intravenous
  Other Names: Sarclisa

SUMMARY:
Primary Objective:

To evaluate the pharmacokinetics (PK) of isatuximab.

Secondary Objectives:

* To evaluate the safety and tolerability of isatuximab.
* To assess the preliminary antitumor effect of isatuximab.
* To evaluate the immunogenicity of isatuximab.

DETAILED DESCRIPTION:
The duration of the study for an individual patient will include a screening period of up to 21 days, a treatment period of repeated 28-day cycles, and a follow-up period. End of treatment visit will be done at 30 (±7) days after last treatment.

ELIGIBILITY:
Inclusion criteria:

* Known diagnosis of symptomatic multiple myeloma.
* At least 2 prior lines of therapies which must include treatment with at least 1 of an immunomodulatory drug (IMiD) or a proteasome inhibitor (PI). The patients must have received an IMiD or a PI for ≥2 cycles or ≥2 months of treatment.
* Patients must have been responsive to at least 1 prior line of therapy (minimal response or better).
* Refractory to the most recently received IMiD or PI included therapy (ie, patients must have progressed during or within 60 days of completion of treatment with IMiD or PI). For patients who have received more than 1 type of IMiD or PI, their disease must be refractory to the most recent one.
* Measurable disease defined as at least 1 of the following:

  * Serum M-protein ≥0.5 g/dL (≥5 g/L);
  * Urine M-protein ≥200 mg/24 hours.
* Written informed consent.

Exclusion criteria:

* <18 years old.
* Eastern Cooperative Oncology Group (ECOG) performance status >2.
* Life expectancy of less than 3 months.
* Pretreated with any anticluster of differentiation (CD) 38 agent.
* Concurrent plasma cell leukemia.
* Known amyloidosis.
* Disease measurable only by serum free light chain (FLC) analysis.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-10-22 (Actual); Primary Completion 2020-09-06 (Actual); Study Completion 2023-08-25 (Actual)

PRIMARY OUTCOMES:
Assessment of PK: Cmax | Cycle 1, up to 168 hours after start of infusion
  To evaluate the maximum observed concentration (Cmax)
Assessment of PK: tmax | Cycle 1, up to 168 hours after start of infusion
  To evaluate the time to reach Cmax (tmax)
Assessment of PK: AUC0-168h | Cycle 1, up to 168 hours after start of infusion
  To evaluate area under the plasma concentration versus time curve over the dosing interval (AUC0-168h)
Assessment of PK: Ceoi | Cycle 1 Day 1, Cycle 2 Day 1, Cycle 4 Day 1; Cycle duration is 28 days
  To evaluate the concentration observed at the end of an IV infusion (Ceoi)
Assessment of PK: Ctrough | Up to approximately 40 weeks (Cycle 10)
  To evaluate concentration observed just before investigational medicinal product (IMP) administration during repeated dosing (Ctrough)

SECONDARY OUTCOMES:
Adverse Events | Up to 30 days after the last IMP administration
  Treatment Emergent Adverse Events (TEAEs)/Serious Adverse Events (SAE) based on standard and systematic assessment including infusion associated reactions (IARs), laboratory test abnormalities, vital signs and ECOG performance status
Anti-tumor activity: Overall response (ORR) | Up to 12 months after last patient treated
  Proportion of patients achieving: stringent complete response (sCR), complete response (CR), very good partial response (VGPR), or partial response (PR) according to International Myeloma Working Group (IMWG 2016) criteria
Anti-Tumor Activity: Duration of response (DOR) | Up to 12 months after last patient treated
  Time from the date of the first determined response to the date of subsequent determined progressive disease or death, whichever happens earlier
Anti-Tumor Activity: Time to progression (TTP) | Up to 12 months after last patient treated
  Time interval from the date of first IMP administration to the date of the first assessed disease progression using IMWG criteria
Anti-Tumor Activity: Progression free survival (PFS) | Up to 12 months after last patient treated
  Time interval from the date of first IMP administration to the date of the first documentation of disease progression or death due to any cause, whichever comes first
Anti-Tumor Activity: Overall survival (OS) | Up to 12 months after last patient treated
  Time interval from the date of first IMP administration to death due to any cause
Immunogenicity | Up to 13 months (10 cycles + 3 months) after last patient treated
  To evaluate the presence of antidrug antibodies (ADA) to isatuximab

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (3):
- China (3):
  - Investigational Site Number 1560003, Beijing
  - Investigational Site Number 1560002, Nanjing
  - Investigational Site Number 1560001, Tianjin

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Sun M, Jing H, Qu X, Dong F, Li Y, Feng Z, Ziti-Ljajic S, Semiond D, Li L, Qi J, Qiu L. Phase 1 study of isatuximab monotherapy in Chinese patients with relapsed/refractory multiple myeloma. Sci Rep. 2024 Nov 11;14(1):27550. doi: 10.1038/s41598-024-59186-1. PMID 39528489